CLINICAL TRIAL: NCT00545142
Title: Multi-center, Single Arm, Open Phase IV Clinical Trial to Evaluate the Efficacy and Safety of Co-administration of Abilify With Depakote in the 6-week Treatment of Acute Mania in Patients With Bipolar Disorder
Brief Title: Abilify in Bipolar Disorder for 6 Weeks Treatment Effectiveness
Acronym: SMART-A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Jeong, Yonghui, Korea Otsuka Pharmaceutical Co.,Ltd.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 031-KOB-0701
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2010-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Abilify(Aripiprazole) — co-administration of Abilify with Depakote in the 6-week treatment of acute mania in patients with bipolar disorder
Drug: Depakote(Divalproate) — co-administration of Abilify with Depakote in the 6-week treatment of acute mania in patients with bipolar disorder

SUMMARY:
To demonstrate the efficacy and safety of co-administration of Abilify(aripiprazole) with Depakote(divalproate) in the acute phase of 6-week treatment of acute mania in patients with bipolar disorder.

DETAILED DESCRIPTION:
Further study details as provided by Korea OIAA

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Mania or mixed episode of Bipolar disorder Bipolar disorder, mania or mixed episode according to DSM-IV
2. The periods of mania or mixed episode should be within 3 months, and YMRS score at enrollment be more than 20.
3. Male and female between the age of 18 and 65 (In case of child-bearing women, negative pregnancy test results should be confirmed before the administration of the investigational drug and appropriate contraception be used. Pregnant and breast-feeding women cannot be included)
4. Patients who can consent to participate in this clinical trial
5. Patients who understand this trial and comply with all protocol requirements

Exclusion Criteria:

1. Patients with the following clinical symptoms diagnosed using DSM-IV:

   * Delirium, dementia, amnestic or other cognitive disorders
   * Schizophrenia or schizoaffective disorder
2. Patients who do not respond to clozapine
3. Patients who are expected to require the administration of prohibited concomitant drugs during the clinical trial period
4. Patients diagnosed with substance-related disorder according to DSM-IV within the past 3 months (abuse, intoxication, dependency and/or withdrawal symptoms). The abuse of benzodiazepines is included with the exception of caffeine or nicotine.
5. Patients known to have allergy or hypersensitivity reaction to Ablify(aripiprazole) or other quinolinones
6. Patients at high risk of suicide attempt or with the history of murder or mental status test
7. Patients with the history of neuroleptic malignant syndrome
8. Patients with the past history which may cause serious adverse events that can affect the safety or efficacy evaluation during the clinical trial period
9. Patients with vital sign or ECG results in the clinically significant abnormal laboratory test Patients with clinically significantly abnormal laboratory results, vital sign or ECG results
10. Pregnant women or child-bearing women who do not or cannot use appropriate contraception
11. Patients given psychotropic medications (except benzodiazepines) one day before baseline visit
12. Patients treated with Fluoxetine for the last 4 weeks
13. Patients who participated in clinical trials with other investigational drugs for the last one month
14. Patients with the history of convulsive disorder
15. Patients with the history of more than 4 mood episodes each year (rapid cycling) during the last 2 years prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes in the YMRS total score from baseline to the end of 6-week study | Throughout the study

SECONDARY OUTCOMES:
Changes in YMRS total scores from baseline to the end of 6-week study | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Won-Myong Bahk, MD, Principal Investigator — St Mary's Hospital, London
Locations (1):
- St. Mary's hospital, Seoul, South Korea